CLINICAL TRIAL: NCT06826950
Title: The Impact of Comprehensive Pharmaceutical Services on Medication Safety in Gynaecological Oncology Chemotherapy Patients
Brief Title: Impact of Pharmacy Services on Gynaecology Chemotherapy Safety
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Zhiqi Zhang, Pharmacist, Peking University First Hospital
Other Study IDs: 2024Y511-002; 2024SF58 (Other Grant/Funding Number: Peking University First Hospital, China)
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Neoplasms; Gynaecological Oncology
Keywords: Pharmaceutical Services; Neoplasms; Chemotherapy; Gynaecological Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group
  Interventions: Other: Routine pharmaceutical services
- Intervention group
  Interventions: Other: comprehensive pharmaceutical care

INTERVENTIONS:
Other: comprehensive pharmaceutical care — The intervention group received comprehensive pharmaceutical care in addition to standard care. For first-cycle patients, oncology pharmacists conducted patient education, informing them about potential chemotherapy-induced adverse reactions and corresponding management strategies. Patients were instructed on the proper use of antiemetic medications, the recommended frequency of blood routine tests, and the appropriate timing, dosing, and administration of granulocyte colony-stimulating factor (G-CSF) and thrombopoietic agents. A QR code for oncology pharmacist consultation was provided to enable patients to seek advice on medication-related issues encountered outside the hospital.
  Groups: Intervention group
Other: Routine pharmaceutical services — The control group received standard care: After the doctor issues the chemotherapy order, the oncology pharmacist only reviews the order to ensure that the chemotherapy regimen and pretreatment regimen during the study are consistent with those of the experimental group. No other interventions are performed.
  Groups: Control group

SUMMARY:
What was studied? We wanted to see whether having pharmacists closely involved in cancer care improves medication safety and reduces severe side effects for patients with gynecologic cancers (like ovarian or uterine cancer) during chemotherapy.

How was the study done?

Who participated? Patients receiving chemotherapy at Peking University First Hospital's Gynecologic Oncology Ward (September 2022-September 2024).

Two groups compared:

Standard care group: Pharmacists provided routine pharmaceutical services.

Full pharmacy care group: Pharmacists provided ongoing support, including:

Checking medications for safety.

Teaching patients how to manage side effects.

Answering questions about drugs.

Helping manage reactions like nausea or low white blood cells.

What was measured? Severe side effects (e.g., extreme nausea, appetite loss), how well doctors prescribed and monitored medications to boost white blood cells, and unplanned hospital stays.

Key findings:

Patients with full pharmacy care had:

Fewer severe side effects: Less extreme nausea, appetite loss, and dangerously low white blood cell counts.

Better management of blood cell-boosting medications: Doctors followed guidelines more closely, and patients received proper monitoring.

Fewer unplanned hospital visits: Likely due to better side effect prevention and early intervention.

Why does this matter?

For patients: Pharmacist support during chemotherapy may help you avoid severe side effects and reduce unexpected hospital stays.

For families: Knowing pharmacists are actively involved can provide reassurance about your loved one's medication safety.

For healthcare teams: Structured pharmacist collaboration improves adherence to treatment guidelines and patient outcomes.

Takeaway:

Full pharmacy care throughout chemotherapy helps protect patients' safety, reduces severe reactions, and supports smoother treatment journeys.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with gynaecologic malignancies such as ovarian cancer, cervical cancer, endometrial cancer, or gestational trophoblastic tumours.
* Patients who received one of the following chemotherapy regimens: taxane monotherapy or combination therapy, anthracycline monotherapy or combination therapy, platinum-based monotherapy or combination therapy. These chemotherapy regimens could be combined with targeted therapy or immunotherapy.

Exclusion Criteria:

* Patients treated with chemotherapy regimens outside those specified in the inclusion criteria.
* Patients who received only targeted therapy, immunotherapy, endocrine therapy, bone-modifying therapy, or combinations of these treatments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer is a disease that occurs exclusively in individuals of the female biological sex (i.e., those who have ovaries). Therefore, eligibility to participate in research is typically based on **biological sex**, rather than **gender identity**. This means that even if a person's gender identity is not female (such as transgender men or non-binary individuals), they are still eligible to participate in ovarian cancer research as long as they have ovaries.
Study Population: Patients with gynaecological tumours receiving chemotherapy at our hospital
Sampling Method: Non-Probability Sample
Enrollment: 629 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Degree of myelosuppression | From enrollment to the end of treatment at 3 weeks

SECONDARY OUTCOMES:
Degree of adverse gastrointestinal reactions | From enrollment to the end of treatment at 3 weeks
Readmission rate | From enrollment to the end of treatment at 3 weeks

OTHER OUTCOMES:
Chemotherapy-related adverse reactions | From enrollment to the end of treatment at 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Hospital patient data needs to be kept confidential